CLINICAL TRIAL: NCT03090646
Title: Use of Financial Incentives to Increase Live Kidney Donor Follow-up Compliance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Living Legacy Foundation (Unknown); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00126158
Record Dates: First submitted 2017-03-02; First posted 2017-03-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Living Donors; Nephrectomy; Kidney
Keywords: social behavioral; living donor kidney transplant; follow-up; health utilization; incentives

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, nonblinded, two-arm, superiority trial with a 1:1 allocation ratio. Participants allocated to the intervention arm will receive up to three gift cards to a major online retailer in the mail after completion of the required 6-month, 1-year, and 2-year follow-up activities. Participants will be followed for the federally-mandated 2-year follow-up period.
Who Masked: Outcomes Assessor
Masking Description: An analyst on the Johns Hopkins University (JHU) study team (blind to group allocations) will use Stata 15 multiprocessor (MP) for Linux (College Station, Texas, USA) to generate a list of sequential group assignments. This list will be used to create sequentially numbered, sealed, opaque envelopes that will be used to allocate participants to the control or intervention arms. Study personnel who create the sealed envelopes will not be involved in patient recruitment. Study personnel who conduct recruitment will not be permitted to view the list of sequential group assignment, and the envelopes will not be opened until after patients consent to participate. Therefore, group allocation will be concealed to both participants and recruiters until after study enrollment.
  The study is not blinded to providers, patients, or study personnel conducting data collection, but will be blinded to outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants in the control arm will be instructed to attend required follow-up as is standard of care, but will not receive a financial incentive.
- Financial Incentive (Experimental): Up to three gift cards to a major online retailer will be mailed to participants assigned to the intervention arm after complete (i.e. all components addressed) and timely (i.e. within the policy-defined follow-up period) submission of follow-up data at each 6-month, 1-year, and 2-year follow-up visit.
  Interventions: Other: Financial Incentive

INTERVENTIONS:
Other: Financial Incentive — Up to three gift cards to a major online retailer.
  Other Names: Behavioral
  Arms: Financial Incentive

SUMMARY:
This study evaluates whether using small financial incentives increases patient compliance with nationally-mandated living kidney donor follow-up at 6-months, 1-year, and 2-years after donation. Half of participants will receive a financial incentive (mailed gift card) after completing required follow-up activities (brief questionnaire and lab draw), while the other half will be asked to complete the required follow-up activities but will not receive a financial incentive (current standard of care).

DETAILED DESCRIPTION:
Living kidney donors account for nearly a third of kidney transplants performed in the United States each year. While donor nephrectomy poses minimal post-surgical risk, donors face a small but measurable increase in the risk of developing kidney failure and other chronic diseases (including hypertension, chronic kidney disease, and diabetes) in the long-term. Routine screening presents an opportunity for the early detection and management of chronic conditions.

Transplant hospital reporting requirements mandate the submission of laboratory and clinical data at 6-months, 1-year, and 2-years after kidney donation, but less than 50% of hospitals are able to comply. Transplant hospitals commonly cite barriers such as donor inconvenience, direct and indirect costs to donors, donors not wanting to return to the program, and the burden of data collection. Tools to improve donor engagement and strategies that mitigate patient and administrative burden are needed.

Financial incentives have been employed in many realms of healthcare to change health-related behaviors. Financial incentives include a variety of rewards that have an economic value for the recipient, including cash payments, coupons, goods, and services, and have been shown to positively influence both simple (i.e. accomplished through a single action) and complex (i.e. accomplished repeatedly over a period of time, often involving sustained lifestyle modifications) health-related behaviors. However, prior work suggests that the effectiveness of financial incentives in achieving health behavior often varies based on the characteristics of the population and health behavior of interest and may decrease over time.

Given that patient-level factors are commonly cited by transplant hospitals as barriers to compliance with federally-mandated donor follow-up thresholds, financial incentives might be a valuable tool to promote patient engagement in post donation monitoring efforts. However, given the uncertainty in the literature, a randomized controlled trial is necessary to evaluate the effectiveness of using financial incentivization to promote patient compliance with follow-up care in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Have undergone live donor nephrectomy at the Johns Hopkins Hospital Comprehensive Transplant Center (MDJH) or the University of Maryland Medical Center Transplant Center (MDUM).

Exclusion Criteria:

* International live kidney donors
* Non-English speaking live kidney donors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient Compliance with Follow-Up | 2 years
  Rate of policy-defined complete (all components addressed) and timely (within 60 days before or after the 6-month, 1-year, or 2-year post donation date; i.e. 120-day period) submission of data at 6-month, 1-year, and 2-year follow-up visits (assessed separately for each follow-up time point and as a composite outcome over the study period).

SECONDARY OUTCOMES:
Hospital compliance with Reporting Requirements | 2 years
  Transplant hospital-level compliance with the Organ Procurement and Transplantation Network (OPTN) reporting requirements (submission of clinical data for 80% and laboratory data for 75% of donors) at each visit (assessed separately for each follow-up time point and as a composite outcome over the study period).

OTHER OUTCOMES:
Logistical Challenges of Intervention Implementation | 2 years
  Data related to potential logistical challenges of implementing the intervention (e.g., number of mailing attempts necessary, failed delivery attempts, incorrect or out-of-date contact information, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Warren, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Maryland Medical Center Transplant Center, Baltimore, Maryland
  - The Johns Hopkins Hospital Comprehensive Transplant Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boudville N, Prasad GV, Knoll G, Muirhead N, Thiessen-Philbrook H, Yang RC, Rosas-Arellano MP, Housawi A, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Meta-analysis: risk for hypertension in living kidney donors. Ann Intern Med. 2006 Aug 1;145(3):185-96. doi: 10.7326/0003-4819-145-3-200608010-00006. PMID 16880460
- [Background] Muzaale AD, Massie AB, Wang MC, Montgomery RA, McBride MA, Wainright JL, Segev DL. Risk of end-stage renal disease following live kidney donation. JAMA. 2014 Feb 12;311(6):579-86. doi: 10.1001/jama.2013.285141. PMID 24519297
- [Background] Schold JD, Buccini LD, Rodrigue JR, Mandelbrot D, Goldfarb DA, Flechner SM, Kayler LK, Poggio ED. Critical Factors Associated With Missing Follow-Up Data for Living Kidney Donors in the United States. Am J Transplant. 2015 Sep;15(9):2394-403. doi: 10.1111/ajt.13282. Epub 2015 Apr 22. PMID 25902877
- [Background] Brown RS Jr, Higgins R, Pruett TL. The evolution and direction of OPTN oversight of live organ donation and transplantation in the United States. Am J Transplant. 2009 Jan;9(1):31-4. doi: 10.1111/j.1600-6143.2008.02433.x. Epub 2008 Oct 6. PMID 18853948
- [Background] Klein AS, Messersmith EE, Ratner LE, Kochik R, Baliga PK, Ojo AO. Organ donation and utilization in the United States, 1999-2008. Am J Transplant. 2010 Apr;10(4 Pt 2):973-86. doi: 10.1111/j.1600-6143.2009.03008.x. PMID 20420647
- [Background] Waterman AD, Dew MA, Davis CL, McCabe M, Wainright JL, Forland CL, Bolton L, Cooper M. Living-donor follow-up attitudes and practices in U.S. kidney and liver donor programs. Transplantation. 2013 Mar 27;95(6):883-8. doi: 10.1097/TP.0b013e31828279fd. PMID 23388736
- [Background] Living Kidney Donor Follow-Up Conference Writing Group; Leichtman A, Abecassis M, Barr M, Charlton M, Cohen D, Confer D, Cooper M, Danovitch G, Davis C, Delmonico F, Dew MA, Garvey C, Gaston R, Gill J, Gillespie B, Ibrahim H, Jacobs C, Kahn J, Kasiske B, Kim J, Lentine K, Manyalich M, Medina-Pestana J, Merion R, Moxey-Mims M, Odim J, Opelz G, Orlowski J, Rizvi A, Roberts J, Segev DL, Sledge T, Steiner R, Taler S, Textor S, Thiel G, Waterman A, Williams E, Wolfe R, Wynn J, Matas AJ. Living kidney donor follow-up: state-of-the-art and future directions, conference summary and recommendations. Am J Transplant. 2011 Dec;11(12):2561-8. doi: 10.1111/j.1600-6143.2011.03816.x. Epub 2011 Nov 4. PMID 22054039
- [Background] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Brennan TA, Asch DA, Volpp KG. Randomized trial of four financial-incentive programs for smoking cessation. N Engl J Med. 2015 May 28;372(22):2108-17. doi: 10.1056/NEJMoa1414293. Epub 2015 May 13. PMID 25970009
- [Background] Kimmel SE, Troxel AB, Loewenstein G, Brensinger CM, Jaskowiak J, Doshi JA, Laskin M, Volpp K. Randomized trial of lottery-based incentives to improve warfarin adherence. Am Heart J. 2012 Aug;164(2):268-74. doi: 10.1016/j.ahj.2012.05.005. PMID 22877814
- [Background] Haisley E, Volpp KG, Pellathy T, Loewenstein G. The impact of alternative incentive schemes on completion of health risk assessments. Am J Health Promot. 2012 Jan-Feb;26(3):184-8. doi: 10.4278/ajhp.100729-ARB-257. PMID 22208418
- [Derived] Bisen SS, Ishaque T, Thomas AG, Waldram MM, Warren DS, Bannon J, Scalea JR, Segev DL, Garonzik-Wang JM, Massie AB, Levan ML. A Two-Center Randomized Controlled Trial to Assess Financial Incentives for Compliance With Living Kidney Donor Follow-Up in the United States. Clin Transplant. 2025 Dec;39(12):e70401. doi: 10.1111/ctr.70401. PMID 41395879
- [Derived] Levan ML, Waldram MM, DiBrito SR, Thomas AG, Al Ammary F, Ottman S, Bannon J, Brennan DC, Massie AB, Scalea J, Barth RN, Segev DL, Garonzik-Wang JM. Financial incentives versus standard of care to improve patient compliance with live kidney donor follow-up: protocol for a multi-center, parallel-group randomized controlled trial. BMC Nephrol. 2020 Nov 9;21(1):465. doi: 10.1186/s12882-020-02117-9. PMID 33167882